CLINICAL TRIAL: NCT03028753
Title: Accuracy of Bladder Scanners in Post-operative Voiding Trials
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study coordinator left / no other current resources to complete
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11871
Record Dates: First submitted 2017-01-11; First posted 2017-01-23 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All subjects (Experimental): All subjects enrolled in the study will have a back-fill voiding trial performed at the time of catheter removal after urogynecologic surgery.
  Interventions: Device: Bladder scan post void residual; Procedure: Straight catheter post void residual; Procedure: Back fill voiding trial

INTERVENTIONS:
Device: Bladder scan post void residual — After voiding on the commode, all subjects will have a post void residual measured by bladder scanner
  Other Names: Verathon BVI9400 Bladder scanner
Procedure: Straight catheter post void residual — After voiding on the commode and having a post void residual measured by bladder scanner, all subjects will have a post void residual measured by straight catheter performed with usual sterile technique.
Procedure: Back fill voiding trial — Prior to catheter removal, all subjects will undergo a back fill voiding trial. The bag of the foley catheter will be removed and the subjects bladder will be filled with 300cc of normal saline (or as much as they can tolerate). The foley catheter will then be removed and the subject will be asked to void on the commode. The voided volume will be measured.

SUMMARY:
The investigators are trying to determine if using a bladder scanner (type of ultrasound) to check how much urine is left in the bladder is the same as checking that volume with a catheter (tube that goes into your bladder to drain urine). After urogynecologic surgery, the investigators perform a voiding trial. Water is put into the participant's bladder through the catheter (tube draining your bladder). The catheter is then removed and the participant is asked to empty their bladder. After that, the investigators will use the bladder scanner (ultrasound) to see how much urine is left in the participant's bladder. After the ultrasound, the investigators will pass a very small catheter (tube) into the bladder to take out the remaining urine. The investigators will then compare the amount obtained from the catheter to the ultrasound amount. This will also help the investigators to figure out if they need to check how much urine is left in a patient's bladder after the voiding trial.

DETAILED DESCRIPTION:
The primary aim of this study is to determine if bladder scanners are accurate in determining a post-void residual volume (PVR) after Urogynecologic surgery.

The secondary aim of this study is to determine if a post-void residual volume (PVR) measurement is needed after a back-fill voiding trial on Urogynecologic post-op patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Urogynecologic surgery
* Able to consent
* Greater than 18 years old
* Non pregnant

Exclusion Criteria:

* Need for prolonged catheterization
* Unable to consent
* Prisoner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Determine if bladder scanners are accurate in determining a post void residual after urogynecologic surgery | Within 48 hours after surgery

SECONDARY OUTCOMES:
Determine if a post void residual volume measurement is needed after a back-fill voiding trial after urogynecologic surgery | Within 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tanaz Ferzandi, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States